CLINICAL TRIAL: NCT00396318
Title: A Phase III, Open-Label, Single-Arm Study of Tenecteplase for Restoration of Function in Dysfunctional Central Venous Catheters
Brief Title: A Study of Tenecteplase for Restoration of Function in Dysfunctional Central Venous Catheters
Acronym: TROPICS 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N3699g
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-03

CONDITIONS: Dysfunctional Central Venous Access Catheters
Keywords: TNKase; CVA; CVAD; Central venous access catheter
MeSH Terms: interventions — Tenecteplase

ARMS (1):
- Tenecteplase (Experimental)
  Interventions: Drug: tenecteplase

INTERVENTIONS:
Drug: tenecteplase — 2 mL of reconstituted lyophilized tenecteplase instilled into lumen of dysfunctional CVC.
  Patients weighing ≥ 30 kg received 2-mL instillations of tenecteplase (i.e., 2 mg of tenecteplase). Patients weighing < 30 kg received instillations of tenecteplase equal to 110% of the internal lumen volume of the dysfunctional CVC. This dose was rounded to the nearest 0.1 mL and should not have exceeded 2 mL (2 mg).

SUMMARY:
This was a Phase III, open-label, single-arm study that was conducted at 43 centers in the United States and Canada. 251 adult and pediatric patients with dysfunctional central venous catheters (CVCs) were enrolled in the study and treated with one or two doses of tenecteplase.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable, in the opinion of the investigator
* CVC occlusion
* Able to have fluids infused at the volume necessary to instill study drug into the CVC

Exclusion Criteria:

* Able to have 3 mL of blood (patients weighing ≥ 10 kg) or 1 mL of blood (patients weighing < 10 kg) withdrawn from the selected CVC following patient repositioning
* Selected study CVC inserted < 2 days prior to treatment
* Selected study CVC implanted specifically for hemodialysis (HD) or internally coated with any therapeutic agent
* Use of a power injector on the selected study CVC during study drug treatment
* Evidence of mechanical, non-thrombotic occlusion of the selected study CVC (e.g., kink in the catheter or suture constricting the catheter)
* Previously treated in this study or any tenecteplase catheter clearance trial
* Use of any investigational drug or therapy within 28 days prior to treatment
* Use of a fibrinolytic agent (e.g., alteplase, tenecteplase, reteplase, or urokinase) within 24 hours prior to treatment
* Known to be pregnant or breastfeeding at screening
* Known bacteremia or known or suspected infection in the CVC catheter
* Known history of intracranial hemorrhage (within the previous 3 years), intracranial aneurysm, or arteriovenous malformation
* Use of heparin (unfractionated or low molecular weight) or any other anticoagulants within 24 hours prior to treatment, except heparin used for prophylaxis or intermittent or low-dose, continuous infusion of heparin to maintain catheter or vessel patency
* Subjects treated with warfarin only: international normalized ratio (INR) ≥ 3.0 within 7 days prior to Visit 1, or a target INR range that allows for an INR ≥ 3.0
* Initiation of or increase in dose of Plavix® (clopidogrel bisulfate) within 7 days prior to treatment
* At high risk for bleeding events or embolic complications (i.e., recent pulmonary embolus, deep vein thrombosis, endarterectomy, or clinically significant right-to-left shunt) in the opinion of the investigator, or with known condition for which bleeding constitutes a significant hazard
* Known hypersensitivity to tenecteplase or any component of the formulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gillespie, M.D., FASN, Study Director — Quintiles, Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five patients were randomized but not treated, therefore the modified intent to treat (MITT) analysis population was 246.
Groups:
- Tenecteplase: 2 mL tenecteplase administered to dwell for 15 (±5) minutes, after which central venous catheter (CVC) function was assessed. Restoration of CVC function was defined as successful withdrawal of at least 3 mL of blood or fluid and infusion of 5 mL of normal saline in patients weighing ≥ 10 kg, and withdrawal of at least 1 mL of blood or fluid and infusion of 3 mL of normal saline in patients weighing < 10 kg. In CVCs for which function was not restored, study drug was left to dwell for an additional 15 (±5) minutes (30 minutes post-treatment), after which CVC function was assessed as before. In CVCs for which function was not restored, study drug was left to dwell for an additional 90 (±10) minutes (120 minutes post-treatment), after which CVC function was assessed as before. If CVC function was not restored by 120 minutes after Dose 1, Dose 2 was given. Assessment of CVC function was repeated as before, after 15 (±5) minutes and, if needed, after 30 (±5) minutes and 120 (±10) minutes.
Period: At Least One Dose of Tenecteplase (MITT)
Arm/Group | Tenecteplase
Started | 246
Completed | 241
Not Completed | 5
Not completed — Subject withdrew consent | 5
Period: 48- to 96-Hour Follow-Up Period
Arm/Group | Tenecteplase
Started | 246
Completed | 241
Not Completed | 5
Period: 7-Day Post-Treatment Contact
Arm/Group | Tenecteplase
Started | 241
Completed | 240
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tenecteplase
Number analyzed (Participants) | 246
Age Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (26.4)
Age, Customized [Number; unit: participants]
  < 2 years | 10
  ≥ 2 to < 17 years | 62
  ≥ 17 to < 65 years | 111
  ≥ 65 years | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Had Cumulative Restoration Rates of Central Venous Catheter (CVC) Function Following a Single Administration of Tenecteplase
Description: Restoration of CVC function was defined as the successful withdrawal of at least 3 mL of blood or fluid and infusion of 5 mL of normal saline in patients weighing ≥ 10 kg, and withdrawal of at least 1 mL of blood or fluid and infusion of 3 mL of normal saline in patients weighing < 10 kg.
Time Frame: 120 minutes after first dose
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 246
percentage of participants | 72.0 [66.3 to 77.6]

2. Secondary Outcome: Percentage of Patients Who Had Cumulative Restoration Rates of CVC Function Following a Single Administration of Tenecteplase
Description: as for outcome 1
Time Frame: 15 minutes after first dose
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 246
percentage of participants | 29.3 [23.6 to 35.0]

3. Secondary Outcome: Percentage of Patients Who Had Cumulative Restoration Rates of CVC Function Following a Single Administration of Tenecteplase
Description: as for outcome 1
Time Frame: 30 minutes after first dose
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 246
percentage of participants | 53.3 [47.0 to 59.5]

4. Secondary Outcome: Percentage of Patients Who Had Cumulative Restoration Rates of CVC Function Following a Second Administration of Tenecteplase
Description: as for outcome 1
Time Frame: 15 minutes after second dose
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 246
percentage of participants | 76.4 [71.1 to 81.7]

5. Secondary Outcome: Percentage of Patients Who Had Cumulative Restoration Rates of CVC Function Following a Second Administration of Tenecteplase
Description: as for outcome 1
Time Frame: 30 minutes after second dose
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 246
percentage of participants | 78.5 [73.3 to 83.6]

6. Secondary Outcome: Percentage of Patients Who Had Cumulative Restoration Rates of CVC Function Following a Second Administration of Tenecteplase
Description: as for outcome 1
Time Frame: 120 minutes after second dose
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 246
percentage of participants | 81.3 [76.4 to 86.2]

7. Secondary Outcome: Percentage of Patients Who Had Cumulative Restoration Rates of CVC Function Following Administration of One or Two Doses of Tenecteplase
Description: as for outcome 1
Time Frame: Up to 120 minutes post-treatment (Dose 1 or Dose 2)
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 246
percentage of participants
  Through first tenecteplase instillation | 72.0 [66.3 to 77.6]
  Through second tenecteplase instillation | 81.3 [76.4 to 86.2]

8. Secondary Outcome: Percentage of Patients Who Had Cumulative Restoration Rates Restoration Rates of CVC Function at Any Time During the Study and Who Maintained Catheter Patency the Next Time the Catheter Was Assessed, up to 7 Days Following the Last Dose of Tenecteplase
Description: as for outcome 1
Time Frame: Up to 7 days post-treatment
Population: Number of patients (from MITT population) with restored CVC function during the treatment period
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 137
percentage of participants | 81.0 [74.5 to 87.6]

ADVERSE EVENTS:
Time Frame: The period during which SAEs and non-serious AEs were recorded began at the initiation of study treatment and ended at the follow-up visit 48-96 hours after treatment or at subject discontinuation from the study, whichever was earlier.
Description: Modified intent to treat (MITT) population.
  Note: The incidence of each AE/SAE is reported as the number of participants experiencing the event, not the number of occurrences for each AE/SAE.
Arm/Group | Tenecteplase
Serious Adverse Events (participants affected / at risk) | 6/246
Other Adverse Events (participants affected / at risk) | 26/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenecteplase (N=246)
Pyrexia (General disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Catheter Related Infection (Infections and infestations) | 1
Device Malfunction (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenecteplase (N=246)
Neutropenia (Blood and lymphatic system disorders) | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Conjunctivitis (Eye disorders) | 1
Eye Discharge (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 4
Catheter Related Complication (General disorders) | 1
Injection Site Erythema (General disorders) | 1
Pain (General disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Graft Versus Host Disease (Immune system disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 1
Rash Pustular (Infections and infestations) | 1
Streptococcal Bacteraemia (Infections and infestations) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.